CLINICAL TRIAL: NCT00503698
Title: Efficacy and Safety of Somatropin in Adult Patients on Chronic Haemodialysis
Brief Title: The Effect of Somatropin Treatment in Adult Patients on Chronic Dialysis
Acronym: OPPORTUNITY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1630-1453; 2006-004702-56 (EudraCT Number)
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Results first posted 2010-07-13 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Chronic Kidney Disease; End-Stage Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Somatropin (Experimental): Somatropin once daily from week 0 to end of trial
  Interventions: Drug: somatropin
- Placebo (Placebo Comparator): Placebo once daily to end of trial
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: somatropin — 20 mcg/kg/day, injected s.c. (under the skin)
  Arms: Somatropin
Drug: placebo — Placebo injected s.c (under the skin)
  Arms: Placebo

SUMMARY:
This trial is conducted in Africa, Asia, Europe, North and South America and Oceania.

The aim of the trial is to evaluate the effect of somatropin (human growth hormone) on survival (primary end-point; "time to death" and health related quality of life in adult patients on chronic haemodialysis.

DETAILED DESCRIPTION:
The decision to discontinue the trial is not due to safety concerns. The discontinuation is based on an analysis of the significant delay in recruitment of patients which is expected to have a negative impact on the outcome of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Serum albumin as specified in protocol
* Malnourished (based on serum albumin value below 40 g/L, assessed centrally)
* Stable (for 3 months or more) and adequate haemodialysis treatment three months prior to enrolment as defined by Kt/V of more than 1.2

Exclusion Criteria:

* Active malignant disease
* Critical illness requiring treatment in an intensive care unit (ICU)
* Uncontrolled treated/untreated hypertension
* Patients on chronic (more than 3 months) treatment with steroids in doses of more than 10 mg/day prednisolone (or equivalent)
* Patients treated with immunosuppressive agents
* Known Growth Hormone Deficiency
* Patients suffering from any clinically significant disease history in the opinion of the investigator
* Severe illness as defined in the protocol (as judged by the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (332):
- United States (180):
  - Novo Nordisk Investigational Site, Alexander City, Alabama
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Madison, Alabama
  - Novo Nordisk Investigational Site, Mobile, Alabama
  - Novo Nordisk Investigational Site, Montgomery, Alabama
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tempe, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Tuscon, Arizona
  - Novo Nordisk Investigational Site, El Dorado, Arkansas
  - Novo Nordisk Investigational Site, Fort Smith, Arkansas
  - Novo Nordisk Investigational Site, Hot Springs, Arkansas
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, McGehee, Arkansas
  - Novo Nordisk Investigational Site, Paragould, Arkansas
  - Novo Nordisk Investigational Site, Pine Bluff, Arkansas
  - Novo Nordisk Investigational Site, Beverly Hills, California
  - Novo Nordisk Investigational Site, Chula Vista, California
  - Novo Nordisk Investigational Site, Covina, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Glendale, California
  - Novo Nordisk Investigational Site, La Mesa, California
  - Novo Nordisk Investigational Site, Lakewood, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Los Alamitos, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Lynwood, California
  - Novo Nordisk Investigational Site, Merced, California
  - Novo Nordisk Investigational Site, Mission Hills, California
  - Novo Nordisk Investigational Site, Monterey Park, California
  - Novo Nordisk Investigational Site, Mountain View, California
  - Novo Nordisk Investigational Site, Pasadena, California
  - Novo Nordisk Investigational Site, Porterville, California
  - Novo Nordisk Investigational Site, Riverside, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, Torrance, California
  - Novo Nordisk Investigational Site, Vacaville, California
  - Novo Nordisk Investigational Site, Visalia, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Whittier, California
  - Novo Nordisk Investigational Site, Yuba City, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Lakewood, Colorado
  - Novo Nordisk Investigational Site, Middlebury, Connecticut
  - Novo Nordisk Investigational Site, Stamford, Connecticut
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Atlantis, Florida
  - Novo Nordisk Investigational Site, Brandon, Florida
  - Novo Nordisk Investigational Site, Coral Springs, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Naples, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Panama City, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Weston, Florida
  - Novo Nordisk Investigational Site, Zephyrhills, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Augusta, Georgia
  - Novo Nordisk Investigational Site, Macon, Georgia
  - Novo Nordisk Investigational Site, Marietta, Georgia
  - Novo Nordisk Investigational Site, Boise, Idaho
  - Novo Nordisk Investigational Site, Meridian, Idaho
  - Novo Nordisk Investigational Site, Crestwood, Illinois
  - Novo Nordisk Investigational Site, Evergreen Park, Illinois
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, Maywood, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Michigan City, Indiana
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Kansas City, Kansas
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Madisonville, Kentucky
  - Novo Nordisk Investigational Site, Baton Rouge, Louisiana
  - Novo Nordisk Investigational Site, Lafayatte, Louisiana
  - Novo Nordisk Investigational Site, New Iberia, Louisiana
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Shreveport, Louisiana
  - Novo Nordisk Investigational Site, Bethesda, Maryland
  - Novo Nordisk Investigational Site, Easton, Maryland
  - Novo Nordisk Investigational Site, Hagerstown, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Silver Spring, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Brockton, Massachusetts
  - Novo Nordisk Investigational Site, Springfield, Massachusetts
  - Novo Nordisk Investigational Site, Dearborn, Michigan
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Lansing, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Columbus, Mississippi
  - Novo Nordisk Investigational Site, Gulfport, Mississippi
  - Novo Nordisk Investigational Site, Jackson, Mississippi
  - Novo Nordisk Investigational Site, City of Saint Peters, Missouri
  - Novo Nordisk Investigational Site, Saint Ann, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Kearney, Nebraska
  - Novo Nordisk Investigational Site, North Platte, Nebraska
  - Novo Nordisk Investigational Site, Eatontown, New Jersey
  - Novo Nordisk Investigational Site, Livingston, New Jersey
  - Novo Nordisk Investigational Site, Voorhees Township, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, Cooperstown, New York
  - Novo Nordisk Investigational Site, Fresh Meadows, New York
  - Novo Nordisk Investigational Site, Mineola, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Port Washington, New York
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, Rosedale, New York
  - Novo Nordisk Investigational Site, The Bronx, New York
  - Novo Nordisk Investigational Site, Yonkers, New York
  - Novo Nordisk Investigational Site, Durham, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Hamlet, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Xenia, Ohio
  - Novo Nordisk Investigational Site, Bend, Oregon
  - Novo Nordisk Investigational Site, Medford, Oregon
  - Novo Nordisk Investigational Site, Roseburg, Oregon
  - Novo Nordisk Investigational Site, Allentown, Pennsylvania
  - Novo Nordisk Investigational Site, Johnstown, Pennsylvania
  - Novo Nordisk Investigational Site, Lewistown, Pennsylvania
  - Novo Nordisk Investigational Site, Meadville, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Providence, Rhode Island
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Columbia, South Carolina
  - Novo Nordisk Investigational Site, North Charleston, South Carolina
  - Novo Nordisk Investigational Site, Orangeburg, South Carolina
  - Novo Nordisk Investigational Site, Santee, South Carolina
  - Novo Nordisk Investigational Site, Sumter, South Carolina
  - Novo Nordisk Investigational Site, Sioux Falls, South Dakota
  - Novo Nordisk Investigational Site, Clarksville, Tennessee
  - Novo Nordisk Investigational Site, Dyersburg, Tennessee
  - Novo Nordisk Investigational Site, Knoxville, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Killeen, Texas
  - Novo Nordisk Investigational Site, Lubbock, Texas
  - Novo Nordisk Investigational Site, McAllen, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Tyler, Texas
  - Novo Nordisk Investigational Site, Weslaco, Texas
  - Novo Nordisk Investigational Site, Provo, Utah
  - Novo Nordisk Investigational Site, Burlington, Vermont
  - Novo Nordisk Investigational Site, Alexandria, Virginia
  - Novo Nordisk Investigational Site, Charlottesville, Virginia
  - Novo Nordisk Investigational Site, Chesapeake, Virginia
  - Novo Nordisk Investigational Site, Fairfax, Virginia
  - Novo Nordisk Investigational Site, Hampton, Virginia
  - Novo Nordisk Investigational Site, Mechanicsville, Virginia
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Portsmouth, Virginia
  - Novo Nordisk Investigational Site, Salem, Virginia
  - Novo Nordisk Investigational Site, Seattle, Washington
  - Novo Nordisk Investigational Site, Bluefield, West Virginia
  - Novo Nordisk Investigational Site, Glendale, Wisconsin
  - Novo Nordisk Investigational Site, Marshfield, Wisconsin
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
  - Novo Nordisk Investigational Site, Neenah, Wisconsin
  - Novo Nordisk Investigational Site, Oshkosh, Wisconsin
- Argentina (8):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Morón
  - Novo Nordisk Investigational Site, Pergamino
  - Novo Nordisk Investigational Site, San Miguel de Tucumán
  - Novo Nordisk Investigational Site, Sarandí
  - Novo Nordisk Investigational Site, Temperley
- Brazil (8):
  - Novo Nordisk Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Novo Nordisk Investigational Site, Curitiba
  - Novo Nordisk Investigational Site, Fortaleza
  - Novo Nordisk Investigational Site, Jaboatao de Guararapes
  - Novo Nordisk Investigational Site, Porto Alegre
  - Novo Nordisk Investigational Site, São José Rio Preto
  - Novo Nordisk Investigational Site, São Paulo
  - Novo Nordisk Investigational Site, Sorocaba
- Canada (11):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Greenfield Park
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Peterborough
  - Novo Nordisk Investigational Site, Regina
  - Novo Nordisk Investigational Site, Saskatoon
  - Novo Nordisk Investigational Site, Scarborough
  - Novo Nordisk Investigational Site, Thunder Bay
- China (3):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Nanjing, Jiangsu
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
- Denmark (7):
  - Novo Nordisk Investigational Site, Aalborg
  - Novo Nordisk Investigational Site, Arhus N
  - Novo Nordisk Investigational Site, Copenhagen
  - Novo Nordisk Investigational Site, Herlev
  - Novo Nordisk Investigational Site, Hilleroed
  - Novo Nordisk Investigational Site, Holbæk
  - Novo Nordisk Investigational Site, Odense
- France (13):
  - Novo Nordisk Investigational Site, Béziers
  - Novo Nordisk Investigational Site, Bordeaux
  - Novo Nordisk Investigational Site, Cherbourt-Octeville
  - Novo Nordisk Investigational Site, Clermont-Ferrand
  - Novo Nordisk Investigational Site, Dunkirk
  - Novo Nordisk Investigational Site, Lyon
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Muret
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Poissy
  - Novo Nordisk Investigational Site, Trappes
  - Novo Nordisk Investigational Site, Vichy
- Germany (25):
  - Novo Nordisk Investigational Site, Aschaffenburg
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Bamberg
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Bernkastel-Kues
  - Novo Nordisk Investigational Site, Bottrop
  - Novo Nordisk Investigational Site, Dormagen
  - Novo Nordisk Investigational Site, Düsseldorf
  - Novo Nordisk Investigational Site, Elsenfeld
  - Novo Nordisk Investigational Site, Fürstenzell
  - Novo Nordisk Investigational Site, Gütersloh
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hanover
  - Novo Nordisk Investigational Site, Heilbronn
  - Novo Nordisk Investigational Site, Kiel
  - Novo Nordisk Investigational Site, Krefeld
  - Novo Nordisk Investigational Site, Limburg an der Lahn
  - Novo Nordisk Investigational Site, Lüdenscheid
  - Novo Nordisk Investigational Site, Mettmann
  - Novo Nordisk Investigational Site, Minden
  - Novo Nordisk Investigational Site, Nettetal
  - Novo Nordisk Investigational Site, Passau
  - Novo Nordisk Investigational Site, Schweinfurt
  - Novo Nordisk Investigational Site, Straubing
  - Novo Nordisk Investigational Site, Würzburg
- Hungary (4):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Eger
  - Novo Nordisk Investigational Site, Kecskemét
  - Novo Nordisk Investigational Site, Sopron
- India (3):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Hyderabad
  - Novo Nordisk Investigational Site, Pune
- Israel (7):
  - Novo Nordisk Investigational Site, Ashkelon
  - Novo Nordisk Investigational Site, Hadera
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Rehovot
  - Novo Nordisk Investigational Site, Tzriffin
- Italy (6):
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Brescia
  - Novo Nordisk Investigational Site, Genova
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Modena
  - Novo Nordisk Investigational Site, Pavia
- Poland (14):
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Kraśnik
  - Novo Nordisk Investigational Site, Kwidzyn
  - Novo Nordisk Investigational Site, Myślenice
  - Novo Nordisk Investigational Site, Ostrów Mazowiecka
  - Novo Nordisk Investigational Site, Poznann
  - Novo Nordisk Investigational Site, Puławy
  - Novo Nordisk Investigational Site, Radom
  - Novo Nordisk Investigational Site, Sieradz
  - Novo Nordisk Investigational Site, Sochaczew
  - Novo Nordisk Investigational Site, Słupca
  - Novo Nordisk Investigational Site, Ul Mlynska 5
  - Novo Nordisk Investigational Site, Wejherowo
  - Novo Nordisk Investigational Site, Wroclaw
- Portugal (10):
  - Novo Nordisk Investigational Site, Abrantes
  - Novo Nordisk Investigational Site, Amadora
  - Novo Nordisk Investigational Site, Braga
  - Novo Nordisk Investigational Site, Corroios
  - Novo Nordisk Investigational Site, Entroncamento
  - Novo Nordisk Investigational Site, Evora
  - Novo Nordisk Investigational Site, Setúbal
  - Novo Nordisk Investigational Site, Torres Vedras
  - Novo Nordisk Investigational Site, Villa Franca de Xira
  - Novo Nordisk Investigational Site, Villa Nova de Gaia
- Novo Nordisk Investigational Site, Ponce, Puerto Rico
- Russia (3):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Petrozavodsk
  - Novo Nordisk Investigational Site, Saint Petersburg
- South Africa (2):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Obervatory
- Spain (8):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Burgos
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Granollers
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Santander
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
- Sweden (3):
  - Novo Nordisk Investigational Site, Stockholm
  - Novo Nordisk Investigational Site, Uppsala
  - Novo Nordisk Investigational Site, Värnamo
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Istanbul
- United Kingdom (14):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Londonderry
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Rhyl
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Swansea
  - Novo Nordisk Investigational Site, Wolverhampton

REFERENCES:
- [Result] Kopple JD, Cheung AK, Christiansen JS, Djurhuus CB, El Nahas M, Feldt-Rasmussen B, Lange M, Mitch WE, Wanner C, Wiedemann J, Ikizler TA. OPPORTUNITY: a randomized clinical trial of growth hormone on outcome in hemodialysis patients. Clin J Am Soc Nephrol. 2008 Nov;3(6):1741-51. doi: 10.2215/CJN.02760608. PMID 18945992
- [Result] Raff AC, Meyer TW, Hostetter TH. New insights into uremic toxicity. Curr Opin Nephrol Hypertens. 2008 Nov;17(6):560-5. doi: 10.1097/MNH.0b013e32830f45b6. PMID 18941347
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 202 sites in 17 countries: United States, Canada, United Kingdom, Sweden, Denmark, France, Germany, Poland, Hungary, Spain, Portugal, Turkey, Israel, Argentina, Brazil, Russia, South Africa. Italy planned to participate but never randomised any subjects.
Pre-assignment Details: Subjects who were malnourished (based on serum albumin value below 40 g/L, assessed centrally) and had received adequate haemodialysis treatment for more than three months at time of trial entry, were eligible.
Groups:
- Somatropin: Somatropin 20 mcg/kg once daily, week 0 to end of trial
- Placebo: Placebo once daily, week 0 to end of trial
Period: Overall Study
Arm/Group | Somatropin | Placebo
Started | 357 (Randomised) | 355 (Randomised)
Exposed to Trial Drug | 346 (11 subjects randomised but not exposed to trial drug. Subjects not included in full analysis set.) | 349 (6 subjects randomised but not exposed to trial drug. Subjects not included in full analysis set.)
Completed | 0 (Trial prematurely terminated) | 0 (Trial prematurely terminated)
Not Completed | 357 | 355
Not completed — Protocol Violation | 5 | 6
Not completed — Adverse Event | 52 | 41
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 3 | 4
Not completed — Trial terminated | 216 | 253
Not completed — End hemodialysis due to renal transplant | 10 | 4
Not completed — Pregnancy/intention to become pregnant | 1 | 0
Not completed — Any condition in exclusion criteria | 4 | 6
Not completed — Switch to peritoneal or home dialysis | 2 | 2
Not completed — Move to nonparticipating dialysis center | 2 | 1
Not completed — Critically ill | 2 | 0
Not completed — Unclassified | 48 | 32
Not completed — Not exposed to trial drug | 11 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Somatropin | Placebo | Total
Number analyzed (Participants) | 346 | 349 | 695
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (13.5) | 61.0 (14.2) | 61.6 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 139 | 314
  Male | 171 | 210 | 381
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 66 | 121
  Not Hispanic or Latino | 286 | 279 | 565
  Unknown or Not Reported | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 114 | 113 | 227
  White | 205 | 213 | 418
  More than one race | 14 | 17 | 31
  Unknown or Not Reported | 3 | 0 | 3
Diabetes [Number; unit: participants]
  Type 1 diabetes mellitus | 12 | 16 | 28
  Type 2 diabetes mellitus | 161 | 150 | 311
  Not Diabetic | 173 | 183 | 356
BMI [Mean (Standard Deviation); unit: kg/m2] — BMI = Body Mass Index
  kg/m2 | 28.9 (8.6) | 28.4 (8.0) | 28.7 (8.3)
Duration of Diabetes [Median (Full Range); unit: years] — Number of years since diagnosis
  years | 17.5 [1.6 to 63.6] | 20.3 [1.2 to 58.5] | 18.4 [1.2 to 63.6]
Duration of Dialysis [Median (Full Range); unit: years] — Number of years in dialysis
  years | 2.9 [0.2 to 27.1] | 2.9 [0.3 to 34.6] | 2.9 [0.2 to 34.6]
Height [Mean (Standard Deviation); unit: cm] | 167.1 (11.2) | 168.1 (10.4) | 167.6 (10.8)
Weight [Mean (Standard Deviation); unit: kg] | 80.6 (24.3) | 80.6 (25.0) | 80.6 (24.6)

OUTCOME MEASURES:

1. Primary Outcome: Mortality - Time to All-cause Death
Description: Time to all-cause death. Statistical analysis is based on all available information from week 0 to trial termination. Summary data illustrates percentage (%) participants dead estimated using Kaplan-Meier. Summary data illustrates mortality until 52 weeks, because very few subjects had trial time longer than 52 weeks. Due to early trial termination, median trial time was 17.4 weeks.
Time Frame: week 0, trial termination
Population: FAS (full analysis set) is all subjects exposed to at least one dose of trial drug. Due to the early termination of this trial, observations from end of trial visit are substituted for week 104 visit (end of trial as per protocol).
Measure: Number; unit: percentage of participants
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 346 | 349
percentage of participants
  Baseline (week 0) | 0 (NA) | 0 (NA)
  Week 26 | 8 | 8
  Week 44 | 13 | 17
  Week 52 | 29 | 23
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Superiority or Other; p = 0.91, Regression, Cox; Time to all-cause death analysed using stratified Cox regression model with treatment and sex as fixed factors, age and time in dialysis as covariates; Cox Proportional Hazard = 0.97, 95% CI 2-sided [0.60 to 1.57]

2. Secondary Outcome: Morbidity - Time From Randomisation to Next Cardiovascular Event (Defined as Composite of All-cause Mortality, Non-fatal Myocardial Infarction, Stroke, Cardiac Insufficiency and Other Thrombo-embolic Event)
Description: Morbidity - time from week 0 to next cardiovascular event (composite of all-cause mortality and cardiovascular events defined as adjudicated medical event of special interest and categorised as myocardial infarctions, cardiac insufficiencies, strokes or other thrombo-embolic events). Statistical analysis is based on all available information from week 0 to trial termination. Summary data illustrates percentage (%) participants with events estimated using Kaplan-Meier. Summary data illustrates morbidity until 52 weeks, because very few subjects had trial time longer than 52 weeks.
Time Frame: week 0, trial termination
Population: FAS (full analysis set) is all subjects exposed to at least one dose of trial drug. Due to the early termination of this trial, observations from end of trial visit are substituted for week 104 (end of trial per protocol).
Measure: Number; unit: percentage of participants
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 346 | 349
percentage of participants
  Baseline (week 0) | 0 (0) | 0 (0)
  Week 26 | 12 | 17
  Week 40 | 18 | 23
  Week 52 | 31 | 24
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Superiority or Other; p = 0.4977, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Cox Proportional Hazard = 0.88, 95% CI 2-sided [0.60 to 1.28]

3. Secondary Outcome: Morbidity - Number of Hospitalisations, in Addition to Normal Dialysis Procedures
Description: The number of times that the patient was hospitalised in addition to hospitalisation for normal dialysis procedures measured from week 0 (randomisation) to the time the trial was terminated.
Time Frame: week 0, trial termination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hospitalisations
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 346 | 349
hospitalisations | 0.5 (0.9) | 0.5 (1.0)
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Superiority or Other; p = 0.4409, Negative binomial regression; Rate ratio = 1.13, 95% CI 2-sided [0.83 to 1.53]

4. Secondary Outcome: Mortality - Two-year Mortality Rate
Time Frame: week 0, trial termination
Population: No analysis was done since the trial was prematurely terminated before week 104 of the trial. Trial was terminated January 16th, 2009.
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Health Related Quality of Life Assessments
Description: Summary from activity of daily living from the Rotterdam Symptom Checklist (RSCL) measuring activity from 1 (active) to 5 (inactive). The Edmonton Symptom Assessment System (ESAS), subjects assess their health in the last 24 hours on a scale from 1 (good health) to 3 (feeling poorly). The EQ-5D is a measure of subjects' health outcome from 0 (death) to 1 (full health). SF-36 (Short Form (36)) covering mental and physicial health is provided in a scale from 0-100 with higher scores indicating greater satisfaction.
Time Frame: week 0, trial termination
Population: FAS (full analysis set) is all subjects exposed to at least one dose of trial drug. Observations from end of trial visit is substitute for week 104. Not all subjects provided 'quality of life' data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 346 | 349
scores on a scale
  RSCL (overall mean), N= 316, 312 | 2.9 (0.9) | 3.0 (0.9)
  ESAS (overall mean), N= 309, 313 | 3.0 (1.9) | 3.0 (2.0)
  EQ-5D (UK overall score), N= 305, 299 | 0.596 (0.310) | 0.597 (0.321)
  SF-36 (overall physical health), N= 318, 315 | 48 (22) | 49 (22)
  SF-36 (overall mental health), N= 318, 315 | 61 (21) | 62 (21)

ADVERSE EVENTS:
Time Frame: The adverse events were collected from July 2007 to January 2009.
Description: The safety analysis set contains all randomised subjects exposed to at least one dose of trial medication.
Arm/Group | Somatropin | Placebo
Serious Adverse Events (participants affected / at risk) | 122/346 | 136/349
Other Adverse Events (participants affected / at risk) | 225/346 | 264/349
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatropin (N=346) | Placebo (N=349)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 7 (9) | 12 (15)
Myocardial infarction (Cardiac disorders) | 4 (4) | 9 (10)
Atrial fibrillation (Cardiac disorders) | 7 (7) | 5 (5)
Cardiac arrest (Cardiac disorders) | 2 (2) | 8 (9)
Coronary artery disease (Cardiac disorders) | 5 (5) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 2 (2)
Angina pectoris (Cardiac disorders) | 3 (3) | 4 (4)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 6 (6)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac asthma (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Electromechanical dissociation (Cardiac disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (6) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 4 (4) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (3)
Multi-organ failure (General disorders) | 2 (2) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Sudden death (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 2 (2) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 10 (11) | 8 (9)
Sepsis (Infections and infestations) | 2 (2) | 7 (8)
Cellulitis (Infections and infestations) | 1 (1) | 5 (5)
Gangrene (Infections and infestations) | 3 (3) | 3 (3)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 4 (4)
Lobar pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Arteriovenous graft site infection (Infections and infestations) | 1 (1) | 3 (3)
Bacteraemia (Infections and infestations) | 1 (1) | 3 (3)
Osteomyelitis (Infections and infestations) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 3 (3) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Staphylococcal infection (Infections and infestations) | 1 (1) | 2 (2)
Arteriovenous fistula site infection (Infections and infestations) | 1 (1) | 1 (1)
Catheter sepsis (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Arteriovenous graft site abscess (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Catheter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Central line infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis viral (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 1 (1)
Graft infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Pathogen resistance (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Subacute endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Underdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound decomposition (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 6 (7) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 7 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Calciphylaxis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carcinoid tumour of the duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 3 (4)
Convulsion (Nervous system disorders) | 2 (2) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Chorea (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium tremens (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (9)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 2 (3)
Deep vein thrombosis (Vascular disorders) | 1 (2) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 2 (2)
Peripheral embolism (Vascular disorders) | 0 (0) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (2)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Exsanguination (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vascular rupture (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatropin (N=346) | Placebo (N=349)
Nausea (Gastrointestinal disorders) | 29 (41) | 36 (39)
Diarrhoea (Gastrointestinal disorders) | 23 (28) | 36 (38)
Vomiting (Gastrointestinal disorders) | 17 (23) | 29 (31)
Asthenia (General disorders) | 9 (11) | 19 (19)
Upper respiratory tract infection (Infections and infestations) | 18 (18) | 11 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (30) | 19 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (23) | 22 (25)
Headache (Nervous system disorders) | 23 (36) | 22 (25)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (24) | 22 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 25 (28)
Hypotension (Vascular disorders) | 24 (33) | 23 (26)

LIMITATIONS AND CAVEATS:
Trial terminated early due to slow recruitment, which largely reduced the power of showing differences. The end of trial visit was used to describe week 104.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.